CLINICAL TRIAL: NCT06687863
Title: Effects of Exercise Training on Neurovascular Control, Endothelial Function, Cognitive Functioning and Genetic Factors in Hypertensive Patients with Obstructive Sleep Apnea Sleep
Brief Title: Effects of Exercise Training and Genetic Factors in Hypertensive Patients with Obstructive Sleep Apnea Sleep
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 5466/22/045
Record Dates: First submitted 2024-02-27; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-02

CONDITIONS: Exercise Training; Genetic Polymorphism
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Masking Description: Data analysis will be carried out by evaluators who do not know the allele of the participant's genetic polymorphism
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OSA training group (Experimental): The training group will be analised compared the effects of exercise on vascular function in different polimorphic aleles.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Includes aerobic exercise, strength training, streching

SUMMARY:
The objective is to investigate the effects of exercise training in hypertensive individuals with obstructive sleep apnea (OSA) in neurovascular control taking into account genetic factors. Seventy-two hypertensive patients with OSA >15 events/hour of sleep revealed by nocturnal polysomnography will be randomized into a control or physical training group. All will be evaluated for the T786 genotypes of the eNOS gene gene. The study will investigate the effect of the exercise program on vascular control in different alleles of the T786 genotypes of the eNOS gene.

DETAILED DESCRIPTION:
Experimental Design. All participants underwent overnight polysomnography study. The apnea-hypopnea index (AHI) will be calculated by total number of respiratory events (apneas and hypopneas) per hour of sleep. Obstructive sleep apnea will be defined as a cessation of respiratory airflow for 10 seconds with thoracoabdominal effort, which was detected by Piezo respiratory effort sensor. Individuals with >70% of obstructive events were defined as individuals with OSA.

Muscle blood flow will be evaluated by pletismography tecnique.

Heart rate and blood pressure. Heart rate (HR) was beat-by-beat continuously measured during the test obtained in a computer-recorded electrocardiographic tracing. Blood pressure (BP) was monitored noninvasively from an automatic leg blood pressure cuff (nondominant leg) using automated oscillometric device. The systolic, diastolic and mean blood pressures will be registered.

Cardiopulmonary Exercise Test. Maximal exercise capacity was determined by means of a maximal progressive cardiopulmonary exercise test Peak VO2 will be defined as the maximum attained VO2 at the end of the exercise period in which the subject could no longer maintain the walk velocity.

ELIGIBILITY:
Inclusion Criteria:

* sedentary,
* Hipertensive patients

Exclusion Criteria:

* Severe cardiovascular, respiratory, renal or severe neuropsychiatric disease

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2028-02-20 (Estimated); Study Completion 2028-02-25 (Estimated)

PRIMARY OUTCOMES:
Genetic polymorphism and obstructive sleep apnea | 4 months of exercise training
  To investigate the effect of exercise training on vascular, sleep parameters, and cognitive function in hypertensive with OSA in different genotypes of the endothelial nitric oxide synthase (eNOS) polymorphism (T786C).

CONTACTS AND LOCATIONS:
Overall Officials: Linda M Ueno-Pardi, Phd, Principal Investigator — USP
Locations (1):
- Linda Massako Ueno Pardi, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No